CLINICAL TRIAL: NCT06138652
Title: Reducing Anxiety Levels Through the Dharma Life App-Based and Mentor-Based Program Targeting Personality Characteristics: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dharma Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00054638
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App (Experimental): Participants completed surveys at baseline and again after 8 weeks. Participants completed app-based games and consultation with a mentor over an 8 week period focused on alleviating anxiety.
  Interventions: Behavioral: App
- Control (No Intervention): Participants completed surveys at baseline and again after 8 weeks.

INTERVENTIONS:
Behavioral: App — Participants completed games on an app and sessions with a mentor focused on alleviating anxiety over 8 weeks.
  Arms: App

SUMMARY:
The purpose of this study was to examine whether an app- and mentor-based program reduced anxiety among individuals reporting difficulties with anxiety.

For the intervention group, this study involved completing an 8-week program focused on helping participants reach their personality goals. The program involved app-based games, journaling, and completing behavioral challenges. Participants engaged with the study app for approximately 15 minutes per day and spoke with a study mentor weekly for 1 hour. Participants were asked to complete surveys prior to and after the program. The pre-program survey lasted approximately 1 hour, and the post-program survey lasted approximately 30 minutes.

For the control group, this study involved completing surveys. Participants were asked to complete surveys 8 weeks apart. The first batch of surveys lasted approximately 1 hour, and the follow-up surveys lasted approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe anxiety levels based on the BAI and GAD-7

Exclusion Criteria:

* We excluded participants experiencing any of the following self-reported behaviors in the past 6 months: substance abuse, self-harm, harm or destruction of another person or their property, suicidal ideations, and feeling helpless after the death of a loved one

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | Baseline and after 8 weeks
  Self report survey of anxiety symptoms
GAD-7 | Baseline and after 8 weeks
  Self report survey of anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Dharma Life Sciences, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No